CLINICAL TRIAL: NCT04195776
Title: A Phase 1 Open Label Study Evaluating the Distribution of a Tenofovir Douche in Combination With Tap Water Douching and Simulated Receptive Anal Intercourse (DREAM-02)
Brief Title: Evaluating Distribution of a Tenofovir Douche With Tap Water Douching and Simulated Receptive Anal Intercourse
Acronym: DREAM-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); CONRAD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00208338; 1U19AI113127 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: HIV/AIDS; HIV Prevention
Keywords: Tenofovir; Tenofovir douche
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Three TFV Medicated Douche Sequences (Experimental): Once enrolled, participants will complete a baseline sampling session and then three sequences of study product administration, along with sRAI and administration of autologous seminal fluid. Sequence A will be 1 TFV douche followed by sRAI; Sequence B will be one dose of TFV douche followed sRAI then a tap water douche; Sequence C will be 1 tap water douche followed sRAI then by a single dose of TFV douche. There will be a washout period of at least 14 days between sequences. Participants will have sequences administered in clinic or a research unit, followed by imaging and various specimen collections over 8 hours.
  Interventions: Drug: Tenofovir Douche

INTERVENTIONS:
Drug: Tenofovir Douche — 660 mg TFV in 125 mL hypo-osmolar solution
  Other Names: TFV 660 mg in hypo-osmolar solution

SUMMARY:
DREAM-02 is a phase 1, open label study to evaluate different sequences of tap water douching and simulated receptive anal intercourse (sRAI) in the presence of a tenofovir douche designed to confer protection from Human Immunodeficiency Virus (HIV) acquisition. DREAM-02 will assess the safety and pharmacokinetics (PK) of different sequences of administration of tap water (H2O) and rectal tenofovir (TFV) douches to more accurately represent the community practice of commonly using cleansing douches prior to RAI, and occasionally after RAI. DREAM-02 results are essential to gain understanding of Tenofovir diphosphate (TFV-DP) concentrations at various anatomic distances in the colon, and how those concentrations may be modified by sRAI, seminal fluid, and sequence of cleansing tap water douches.

DETAILED DESCRIPTION:
DREAM-02 is proposed as the next step in the development of an on demand, behaviorally-congruent rectal tenofovir (TFV) microbicide to prevent HIV acquisition via unprotected receptive anal intercourse (RAI).

The DREAM Program has previously established that (1) no TFV pro-drug provides significantly superior colon tissue pharmacokinetics in pre-clinical models (mice and macaques), (2) a single rectal TFV douche protects macaques from repeated low dose rectal simian/human immunodeficiency virus (SHIV) challenge and is superior to oral daily dosing of TFV disoproxil fumarate (TDF), (3) it takes only 1-3 hours for a single 125 mL hypotonic rectal douche with a concentration of 5.28 mg/mL of TFV (660 mg total)to exceed by 100-fold the steady-state colon tissue TFV diphosphate (TFV-DP) concentrations associated with >90% protection (83 femtomoles/ million [fmol/106] Mucosal Mononuclear Cells (MMC) in oral daily dosing studies), and (4) DREAM behavioral survey research indicates very common use of one to several rectal douches in series prior to Unprotected Receptive Anal Intercourse (URAI).

DREAM-02 will assess the safety and PK of different sequences of administration of tap water (H2O) and rectal TFV douches to more accurately represent the community practice of commonly using cleansing douches prior to RAI, and occasionally after RAI, based on investigators' DREAM behavioral survey results. DREAM-02 results are essential to gain understanding of TFV-DP concentrations at various distances from the anal verge, and how those concentrations may be modified by sRAI, seminal fluid, and sequence of cleansing tap water douches.

The sequences of douche administration are selected to evaluate the impact of either a TFV rectal douche or H2O douche administered prior to, or following simulated sexual intercourse with ejaculation. The first sequence of administration will replicate administration of the dose that achieved the greatest tissue TFV-DP concentrations in DREAM-01 (660 mg TFV in 125 mL half-normal saline; TFV 5.28 mg/mL), then followed by simulated receptive anal intercourse (sRAI) and administration of autologous seminal fluid via a catheter embedded in an artificial phallus (Sequence A). Sequence B will evaluate the administration of the TFV rectal douche administered prior to sRAI and ejaculation followed by a cleansing H2O douche. Lastly, Sequence C will evaluate the administration of a cleansing H2O douche prior to sRAI and ejaculation followed by the TFV rectal douche.

Investigators hypothesize that douching after sex will increase the distribution of HIV surrogates within the lower GI tract and may lead to a mismatch of drug and HIV surrogate distribution, possibly, reducing rectal douche effectiveness. This information will be essential to the design of phase 2 extended safety studies of investigators' TFV douche, especially with regard to providing guidance for research participants and study counselors. Since DREAM-02 and DREAM-03 will use the same TFV douche product, DREAM-02 will provide data complementary to the 3 dose sequences planned for DREAM-03, and in the first arm of this protocol replicates the same product/conditions as used in the highest dose escalation step of DREAM-01, but with the addition of sRAI and exposure to autologous seminal fluid. Therefore, bridging data from DREAM-01, DREAM-02, and DREAM-03, as well as data from other DREAM Projects will inform the design and labeling of an optimal TFV douche for further clinical testing.

It is anticipated that the study will take approximately six months to complete study enrollment, and that each participant will be in the study for approximately six months from the time of screening.

ELIGIBILITY:
Inclusion Criteria:

* Biologically assigned male gender at birth, 18 years of age or older at screening
* Willing and able to communicate in English
* Willing and able to provide written informed consent to take part in the study
* Willing and able to provide adequate locator information
* Understand and agree to local sexually transmitted infection (STI) reporting requirements
* HIV-1 uninfected at screening as documented by Combo Ag/Ab HIV-1/HIV-2 immunoassay
* Willing to provide a semen sample on multiple occasions
* Wiling to perform simulated RAI with the Coital Dynamic Simulation (CDS) device
* Available to return for all study visits, barring unforeseen circumstances
* Per participant report at screening, a history of consensual RAI
* Per participant report at screening, experience with receiving or self-administering a rectal douche in the context of RAI.
* If the study participant is currently prescribed oral TDF 300 mg/emtricitabine (FTC) 200 mg (Truvada®), or FTC 200 mg/tenofovir alafenamide (TAF) 25 mg (Descovy®) as HIV Pre Exposure Prophylaxis (PrEP), the participant may continue to take oral PrEP as prescribed as long as the participant agrees to adhere to a consistent dosing schedule throughout the study duration.
* Willing to abstain from insertion of anything (drug/medication, penis, object, sex toy, or douche) into the anorectum for 72 hours before and after each research unit study product exposure and 7 days after each flexible sigmoidoscopy with biopsy collection.
* Willing to refrain from ejaculation for a period of 48 hours prior to each semen collection
* Willing to refrain from high daily dose aspirin (>81 mg) and NSAID use for one week before and after each study biopsy visit
* Willing and able to use condoms provided by the study for all RAI for the duration of participation
* Agrees not to participate in other research studies involving drugs and/ or medical devices for the duration of the study

Exclusion Criteria:

* History of chronic Hepatitis B infection, as documented by positive HBsAg at screening
* ≥ Grade 2 laboratory abnormality at baseline as defined by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 - July 2017, and Addendum 3 (Rectal Grading Tables for Use in Microbicide Studies)
* Serum phosphate <2.3 mg/dL
* Significant colorectal symptom(s) as determined by medical history or by participant self-report (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, history of inflammatory bowel disease, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation)
* At screening or within the past 2 months: participant-reported symptoms and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active herpes simplex virus (HSV) lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts. Note that HSV seropositivity with no active genital lesions is not an exclusion criterion. (Note: if an STI apart from HIV is detected, the participant will be referred for treatment. For GC/CT the participant can be retested in 30 days and rescreened once. For syphilis, individuals with a positive screening test, but a non-reactive or low titer rapid plasma reagin (RPR) with a history of adequate treatment, may be enrolled. Individuals testing newly positive for syphilis can be enrolled 30 days after documented treatment)
* History of an underlying clinically significant cardiac arrhythmia or renal disease (including creatinine clearance <60 mL/min using Cockcroft-Gault equation)
* History of significant gastrointestinal bleeding
* Current use of warfarin or heparin or other anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], NSAIDs, or Pradaxa®)
* Use of systemic or anorectal immunomodulatory medications within 4 weeks of enrollment or planned use at any time during study participation
* Per participant report, use of any rectally administered products containing N-9 (including condoms) or investigational products within 4 weeks of enrollment, or planned use of either at any time during study participation
* Known allergic reaction to TFV or other components of the test articles
* Current known HIV-infected partners, or if in the opinion of the investigator, the participant identifies as a commercial sex worker, or has frequent unprotected RAI with partners of unknown HIV status.
* Use of injection or non-injections drugs that in the opinion of the investigator could compromise participant safety or the integrity of the study.
* Symptoms suggestive of acute HIV seroconversion at screening and enrollment
* Participants whose whole body (ED) radiation exposure, per participant report, exceeds 5000 mrem/year
* Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will include individuals biologically assigned male gender at birth.
Enrollment: 6 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Tenofovir Diphosphate (TFV-DP) concentration | Approximately 6 months from the time of enrollment
  Colonic tissue cell TFV-DP concentrations (femtomoles/million cells) will be measured 3 hours after each study douche sequence administration.

SECONDARY OUTCOMES:
Anatomic distribution of radiolabeled Tenofovir douche | Approximately 6 months from the time of enrollment
  Tenofovir douches will be radiolabeled with 111In-diethylenetriaminepentaacetic acid (DTPA) Computed tomography (CT) and single photon emission computed tomography (SPECT) imaging will be used at 1 hour after each TFV douche sequence administration to study the distribution of radiolabeled products. Maximal extent of radiosignal distribution from the anal verge, measured in centimeters (cm), will be estimated for each research participant and paired comparisons made between each dosing sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Nimmagadda, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng R, Fuchs EJ, Nimmagadda S, Rohan LC, Wang L, Bertagnolli LN, Massih S, Caffo BS, Hendrix CW. Anal Sex and Tenofovir Douche Sequence Impacts Colorectal Distribution of HIV Surrogate and Douche: DREAM-02. J Infect Dis. 2025 Sep 15;232(3):588-595. doi: 10.1093/infdis/jiaf286. PMID 40447283